CLINICAL TRIAL: NCT02622763
Title: Safety and Clinical Efficacy Evaluation of Intralesional Administration of Tolerogenic Dendritic Cells in Patients With Refractory Crohn's Disease
Brief Title: Intralesional Tolerogenic Dendritic Cells in Crohn's Disease Treatment
Acronym: TolDecCDintra
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TolDec-CD-intra; 2014-001083-35 (EudraCT Number)
Record Dates: First submitted 2015-12-01; First posted 2015-12-04 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Crohn's Disease
Keywords: Tolerogenic Dendritic Cells
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 millions dose (Experimental): a total of 10 millions tolerogenic dendritic cells
  Interventions: Biological: Tolerogenic Dendritic Cells
- 100 millions dose (Experimental): a total of 100 millions tolerogenic dendritic cells
  Interventions: Biological: Tolerogenic Dendritic Cells

INTERVENTIONS:
Biological: Tolerogenic Dendritic Cells — Intralesional administration

SUMMARY:
Intralesional Tolerogenic Dendritic Cells in Crohn's Disease Treatment.

DETAILED DESCRIPTION:
The main objective is to evaluate the safety and clinical response of intralesional injection of Autologous peripheral blood differentiated adult dendritic cells expanded tolerogenic in patients with refractory Crohn's disease treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Crohn's disease ( Lennard -Jones criteria )
2. Active Crohn's disease in the last six months to the inclusion defined as : CDAI? 220 and endoscopic or radiological criteria of activity
3. Refractory or intolerance to conventional therapy including corticosteroids , immunomodulators and anti-tumor necrosis factor-alpha
4. Presence of visible lesions by endoscopy
5. Acceptance to participate in the study and written informed consent

Exclusion Criteria:

1. No injuries in pre-screening resonance
2. Pregnancy, lactation or women of childbearing age not taking appropriate contraceptive measures
3. Patients HIV + and Hepatitis C Virus + Hepatitis B Virus +
4. Serious concomitant disease:

   * Renal failure with creatinine clearance < 40ml / min
   * Heart disease: congestive heart failure with ejection fraction < 45 % , atrial fibrillation treated with oral anticoagulants, uncontrolled ventricular arrhythmias , pericarditis , pleural effusion with hemodynamic
   * Neoplasms or myelodysplasia
   * Psychiatric disorders including alcohol and drugs
5. Symptoms attributable to fibrotic strictures in Crohn's disease at the discretion of the investigators
6. Diarrhea attributable to " short bowel syndrome"
7. Active infection , including tuberculosis
8. Participation in research studies of new drugs in the 3 months prior to inclusion.
9. Vaccination with live/attenuated germs in the previous 3 months
10. Personal history of cancer (active or complete remission) or known family history of hereditary cancer.
11. Patients in whom , after observation of the state of their veins , these are considered inaccessible and impossible to perform apheresis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | from inclusion up to 12 weeks
Proportion of patients with clinical response defined as a decrease of Crohn 's Disease Activity Index > 100 points | up to 12 weeks

SECONDARY OUTCOMES:
The proportion of patients with clinical response defined as a decrease of Crohn 's Disease Activity Index > 100 points | from baseline to week 12
The proportion of patients in clinical remission defined as Crohn 's Disease Activity Index < 150 points | at week 12
Endoscopic lesions using the Crohn 's Disease Endoscopic Index of Severity ". Endoscopic remission was defined as the absence of ulcers | at baseline and week 12
The evaluation of quality of life will be held by Inflammatory bowel disease questionnaire Immunological endpoints | Change from baseline to week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain